CLINICAL TRIAL: NCT05752448
Title: POSTCARE-O: Survivorship Care for Women Living With Ovarian Cancer
Brief Title: Survivorship Care for Women Living With Ovarian Cancer: (POSTCARE-O)
Acronym: POSTCARE-O
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other); The University of Texas Health Science Center, Houston (Other); University of Texas Southwestern Medical Center (Other); University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Elizabeth A Kvale, Associate Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: H-52939
Record Dates: First submitted 2023-02-22; First posted 2023-03-02 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Neoplasm; Depressive Symptoms; Quality of Life
Keywords: Ovarian Cancer; Survivorship; Cancer Survivor; Depression; Palliative Care; Quality of Life
MeSH Terms: conditions — Ovarian Neoplasms; Depression

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial double blinded
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Will mask all study personnel except care provider who will not be engaged with data interpretation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Group received care Using POSTCare process
  Interventions: Behavioral: POSTCare Survivorship transition process
- Usual Care (No Intervention): Group received usual care

INTERVENTIONS:
Behavioral: POSTCare Survivorship transition process — Survivorship coaching intervention
  Arms: Intervention group

SUMMARY:
This study will enroll 120 women living with ovarian cancer following completion of initial treatment. Our objective is to test an intervention designed to provide support during the survivorship transition for this population, who live with a high degree of morbidity related to the illness and its treatment as well as a high risk of recurrence. Study participants will be randomly assigned to receive survivorship care using the POSTCare-O process or usual care. The primary outcome is quality of life at 12 weeks after intervention.

DETAILED DESCRIPTION:
Study Design We will conduct a 2-arm randomized controlled trial to evaluate the impact of a telehealth delivered survivorship transition care process. Ovarian cancer survivors (120) will be randomly allocated to receive survivorship care either using the POSTCare Process or standard of care. Study design and reporting will be in accordance with the Consolidated Standards of Reporting Trials (CONSORT) checklist. We will use quantitative and qualitative methodologies in a concurrent triangulation mixed methods design utilizing qualitative data to augment our interpretation of quantitative data. Outcomes will be collected at baseline, 12 weeks and 24 weeks, with the primary outcome being quality of life assessment at 12 weeks.

Sample Size We will enroll 120 women completing primary treatment for Stage 2-4 ovarian cancer from 3 urban gynecologic oncology clinics located in the Southern United States. Participants will have received some combination of surgery, chemotherapy, radiation therapy, and biologics. Continued maintenance therapy is not an exclusion factor. Aim 1 proposes to implement a randomized controlled trial (RCT) devised to compare QOL measures among ovarian cancer patient randomized to receive usual care versus the POSTCare survivorship care transition program. The Functional Assessment of Cancer Therapy-Ovarian (FACT-O) QOL survey will be collected at baseline as well as 12 and 24 weeks after the initial course of adjuvant chemotherapy. The primary endpoint will be the 12-week survey. We expect to observe a mean 12-week FACT-O score of 116 with standard deviation of 20 for women receiving usual care. The sample size of N=120 patients provides at least 80% power to detect a 7% increase in the mean FACT-O score for women randomized to the POSTCare survivorship care intervention. This is sufficient to ascertain a minimally important difference of 8 points.

Recruitment and Setting We will recruit participants from Gynecologic Oncology practices at 3 clinic settings in Texas: One safety net practice located in Dallas, one safety net practice located in Houston, and one faculty group practice located in Houston. Cumulatively the sites serve approximately 120 eligible patients per year and ensure a diverse population can be recruited during the 24-month recruitment period. 120 women will be recruited. Sixty participants will be randomly assigned to the intervention group and receive care using the POSTCare Process and 60 will be randomly assigned to the control group. It is anticipated that our study sample will reflect the ethnic and racial diversity of our clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Stage 2-4 ovarian cancer
* Treated with some combination of surgery, chemotherapy, biologics, maintenance therapy
* Within 6 months of completion of initial treatment (continued maintenance therapy okay)
* Able to provide consent in English or Spanish

Exclusion Criteria:

* Admission to hospice at the completion of treatment for ovary cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females at birth have ovaries
Enrollment: 120 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Quality of Life by FACT-O | 12 Weeks
  Quality of life measured by Functional Assessment of Cancer Therapy - Ovarian instrument composite scorecomprised of physical, emotional, functional, social, and disease specific subscales. Scoring range 0 - 152; a higher score indicates better quality of life.

SECONDARY OUTCOMES:
Quality of Life by FACT-O | 24 weeks
  Quality of life measured by Functional Assessment of Cancer Therapy - Ovarian instrument composite scorecomprised of physical, emotional, functional, social, and disease specific subscales. Scoring range 0 - 152; a higher score indicates better quality of life.
Recurrence Fear | 12 and 24 weeks
  Fear of Cancer Recurrence measured by Fear of Cancer Recurrence Inventory Short Form. Range 0-36; higher score indicates higher fear of cancer recurrence.
Depressive Symptom Burden | 12 and 24 weeks
  Depression measured by the Patient Health Questionnaire - 9 . Range 0-27; higher score indicates greater depressive symptom burden.
Symptom Burden | 12 and 24 weeks
  Symptom Burden measured by The M.D. Anderson Symptom Inventory. Range is 1-130; higher score indicates greater symptom burden

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Kvale, MD,MPH, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - UT Southwestern Parkland Health and Hospital System, Dallas, Texas
  - Dan L Duncan Comprehensive Cancer Center at the O'Quinn Medical Tower at Baylor St. Luke's Medical Center, Houston, Texas
  - Harris Health Smith Clinic, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kvale E, Phillips F, Ghosh S, Lea J, Hoppenot C, Costales A, Sunde J, Badr H, Nwogu-Onyemkpa E, Saleem N, Ward R, Balasubramanian B. Survivorship Care for Women Living With Ovarian Cancer: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Feb 9;13:e48069. doi: 10.2196/48069. PMID 38335019